CLINICAL TRIAL: NCT03615950
Title: Effects of Swallowed Corticosteroids on Bone Mineral Density and Growth Velocity in Children With Eosinophilic Esophagitis
Brief Title: Effects of Swallowed Steroids on Bone Density and Growth in Pediatric Eosinophilic Esophagitis
Status: Withdrawn | Type: Observational
Why Stopped: No recruitment
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Collaborators: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: ACHEOEBMD
Record Dates: First submitted 2018-07-24; First posted 2018-08-06 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — Bone Density; Absorptiometry, Photon; Radionuclide Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention Group: 30 Children with eosinophilic esophagitis who are started on swallowed corticosteroids by their clinical provider.
  Interventions: Diagnostic Test: Bone Mineral Density (DEXA) scan; Diagnostic Test: Vitamin D Measurement; Diagnostic Test: Height measurement; Other: Assessment of medication compliance
- Control Group: 30 children, 5-12 years of age, not taking swallowed corticosteroids. Age and sex matched 1:1 with intervention group.
  Interventions: Diagnostic Test: Bone Mineral Density (DEXA) scan; Diagnostic Test: Vitamin D Measurement; Diagnostic Test: Height measurement

INTERVENTIONS:
Diagnostic Test: Bone Mineral Density (DEXA) scan — Radiologic assessment of bone mineral density in the lumbar spine. This will be performed at screening. If abnormal at screening, subjects will not be enrolled. For enrolled subjects, DEXA will be repeated at 12 months.
Diagnostic Test: Vitamin D Measurement — Measurement of 25-hydroxy vitamin D levels through the blood at baseline and 12 months. If low for age, subjects will receive dietary counseling to increase intake to recommended levels. Primary care providers of enrolled subjects will be notified of abnormal results.
Diagnostic Test: Height measurement — Height will be measured at baseline and 12 months.
Other: Assessment of medication compliance — Subjects enrolled in the intervention group will undergo assessment of compliance with swallowed corticosteroids prescribed by their clinical provider. This will be performed at 6 and 12 months.
  Groups: Intervention Group

SUMMARY:
Eosinophilic esophagitis (EoE) is characterized by allergy-driven inflammation of the esophagus leading to a variety of gastrointestinal symptoms and increased healthcare utilization. While considered a rare disease, EoE is rapidly increasing in prevalence in the United States. Treatment options are limited and include dietary modifications with the elimination of suspected food triggers or pharmacological options including proton pump inhibitors (PPIs) and swallowed corticosteroids. Compliance to strict elimination diets is difficult thus many patients elect to use swallowed corticosteroids. Because nearly half of all EoE patients are treated with swallowed corticosteroids there is a growing concern regarding the long-term effects of this class of medication.4

It is known that oral corticosteroids can compromise bone mineral density and growth velocity5-7. Furthermore, there have been multiple studies exploring the relationship between inhaled corticosteroids (ICS) and endocrine effects in asthmatics. While the risk of ICS use is less compared to systemic corticosteroids, higher ICS doses do cause deleterious effects on growth and bone health8-11. Currently, there are no published studies examining the effect of swallowed corticosteroids on bone mineral density or growth velocity in patients with EoE. Given the route of administration, there may be more systemic absorption leading to a higher risk of long-term complications.

The proposed work will address the following specific aims:

Specific Aim 1: Assess effects of swallowed corticosteroids on bone mineral density (primary outcome) in children 5-12 years of age with EoE compared to age matched controls.

Specific Aim 2: Evaluation of the effect of swallowed corticosteroids on growth velocity.

ELIGIBILITY:
Inclusion Criteria:

* Intervention:

  1. Age 5-12 years
  2. Diagnosis of EoE based upon a peak eosinophil count of ≥ 15 eosinophils/high powered field (hpf) on at least one esophageal biopsy while on a minimum of 8 weeks of PPI therapy
  3. Patient/Family has elected to start swallowed corticosteroids for the treatment of EoE with a minimum daily dose of at least 0.5 mg budesonide or 440 mcg fluticasone. The decision to start swallowed corticosteroids will be made based upon the judgement of the provider, potential subject, and family during a clinic visit and will not be part of the research procedures.
* Controls:

  1. Age 5-12 years
  2. Followed in the ACH allergy clinic, but not required to have a diagnosis of EoE
  3. Not treated with swallowed corticosteroids

Exclusion Criteria:

* Intervention and controls:

  1. Non-English speaking
  2. Patients actively taking systemic corticosteroids or previous use of systemic corticosteroids within the past 6 months
  3. Patients actively taking inhaled corticosteroids or prior use of inhaled corticosteroids in the 6 months prior to screening
  4. Current or previous treatment with swallowed corticosteroids for EoE at the time of screening
  5. Osteopenia or osteoporosis on baseline dual energy X-ray absorptiometry (DEXA).

Ages: 5 Years to 12 Years | Sex: All
Age Groups: Child
Gender Based: Yes — Male and Female children, 5-12 years of age are eligible. Controls are age and gender matched to those in the intervention group
Study Population: We will recruit 30 children, ages 5-12 years, with eosinophilic esophagitis (EoE) and 30 age and sex-matched controls from the Arkansas Children's Hospital allergy clinic to participate in this prospective study. Controls will be age- and gender-matched in a 1:1 ratio with EoE subjects but will not be required to have a diagnosis of EoE. Control subjects will not be treated with swallowed corticosteroids.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-02 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Effects of swallowed corticosteroids on bone mineral density | 12 months
  Change in bone mineral density over 1 year while being treated with swallowed corticosteroids compared to age-matched controls

SECONDARY OUTCOMES:
Effects of swallowed corticosteroids on linear growth | 12 months
  Changes in linear growth over 1 year while being treated with swallowed corticosteroids compared to controls

CONTACTS AND LOCATIONS:
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No